CLINICAL TRIAL: NCT00057200
Title: Evaluating Telehealth Home Care for Elderly Veterans With Congestive Heart Failure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NRI 99-345
Record Dates: First submitted 2003-03-27; First posted 2003-03-31 (Estimated); Last update posted 2015-04-07 (Estimated); Status verified 2007-02

CONDITIONS: Heart Failure; Telemedicine
Keywords: Home Care
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Other)
  Interventions: Procedure: Telephone, videophone care

INTERVENTIONS:
Procedure: Telephone, videophone care

SUMMARY:
Congestive heart failure (CHF) is one of the most common reasons for hospitalization in patients aged 65 years and older. Many hospitalizations for CHF are potentially preventable if the warning signs of decompensation are recognized and treated before the situation becomes emergent. Home-based intervention programs have reduced unplanned readmission rates for patients with CHF by up to 50 percent. Using advanced telecommunications technologies it is now possible to provide greatly improved access and availability of services in a more timely and cost effective manner directly to patients� homes. Although telehealth offers a number of theoretical advantages, few empirical studies have compared telehealth to traditional delivery modes, and virtually no studies have compared the effectiveness of alternative telehealth applications.

DETAILED DESCRIPTION:
Background:

Congestive heart failure (CHF) is one of the most common reasons for hospitalization in patients aged 65 years and older. Many hospitalizations for CHF are potentially preventable if the warning signs of decompensation are recognized and treated before the situation becomes emergent. Home-based intervention programs have reduced unplanned readmission rates for patients with CHF by up to 50 percent. Using advanced telecommunications technologies it is now possible to provide greatly improved access and availability of services in a more timely and cost effective manner directly to patients� homes. Although telehealth offers a number of theoretical advantages, few empirical studies have compared telehealth to traditional delivery modes, and virtually no studies have compared the effectiveness of alternative telehealth applications.

Objectives:

The purpose of this study is to compare the effectiveness and resource use of two telehealth interventions to traditional care provided for recently discharged outpatients with CHF. Four hypotheses will be tested. Compared to subjects who receive usual care, subjects who receive telehealth interventions (telephone or interactive video) following discharge will: 1) have lower readmission rates; 2) report improved quality of life, self-efficacy, and satisfaction with care; 3) use fewer resources, including hospital days, urgent care visits, and telephone calls; and 4) have higher survival rates.

Methods:

The study is a randomized controlled clinical trial. We will compare usual care to an intervention delivered by either telephone or interactive video to veterans following discharge from the hospital. A total of 198 subjects will be enrolled over three years. Subjects in the treatment groups (telephone or interactive video) will receive the intervention for 90 days following discharge from the hospital. Data to be collected includes measures of quality of life, self-efficacy, satisfaction, resource use, and mortality.

Status:

Project work is ongoing.

ELIGIBILITY:
Inclusion Criteria:

Patients admitted to the Iowa City VA Medical Center for treatment of congestive heart failure exacerbation. Must be cognitively intact and have a telephone line in the home.

Exclusion Criteria:

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 198 (Estimated)
Dates: Study Completion 2005-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bonnie J. Wakefield, PhD RN, Principal Investigator — Iowa City VA Health Care System, Iowa City, IA
Locations (1):
- Iowa City VA Health Care System, Iowa City, IA, Iowa City, Iowa, United States

REFERENCES:
- [Result] Wakefield BJ, Orris LJ, Holman JE, Russell CL. User perceptions of in-home medication dispensing devices. J Gerontol Nurs. 2008 Jul;34(7):15-25. doi: 10.3928/00989134-20080701-10. PMID 18649820
- [Result] Wakefield BJ, Bylund CL, Holman JE, Ray A, Scherubel M, Kienzle MG, Rosenthal GE. Nurse and patient communication profiles in a home-based telehealth intervention for heart failure management. Patient Educ Couns. 2008 May;71(2):285-92. doi: 10.1016/j.pec.2008.01.006. Epub 2008 Mar 11. PMID 18337049
- [Result] Wakefield BJ, Ward MM, Holman JE, Ray A, Scherubel M, Burns TL, Kienzle MG, Rosenthal GE. Evaluation of home telehealth following hospitalization for heart failure: a randomized trial. Telemed J E Health. 2008 Oct;14(8):753-61. doi: 10.1089/tmj.2007.0131. PMID 18954244
- [Result] Wakefield BJ, Holman JE, Ray A, Scherubel M, Burns TL, Kienzle MG, Rosenthal GE. Outcomes of a home telehealth intervention for patients with heart failure. J Telemed Telecare. 2009;15(1):46-50. doi: 10.1258/jtt.2008.080701. PMID 19139220
- [Result] Darkins A, Ryan P, Kobb R, Foster L, Edmonson E, Wakefield B, Lancaster AE. Care Coordination/Home Telehealth: the systematic implementation of health informatics, home telehealth, and disease management to support the care of veteran patients with chronic conditions. Telemed J E Health. 2008 Dec;14(10):1118-26. doi: 10.1089/tmj.2008.0021. PMID 19119835
- [Result] Wakefield BJ, Holman JE, Ray A, Morse J, Kiensie M. Nurse and patient preferences for telehealth home care. Geriatric Times. 2004 Mar 1; V(2):27-30.
- [Result] Wakefield BJ, Holman JE, Ray A, Morse J, Kienzle MG. Nurse and patient communication via low- and high-bandwidth home telecare systems. J Telemed Telecare. 2004;10(3):156-9. doi: 10.1258/135763304323070805. PMID 15165441